CLINICAL TRIAL: NCT06954961
Title: A Randomized, Parallel-controlled, Open-label, Multicenter Phase III Clinical Study to Compare the Efficacy and Safety of D-0502 With Fulvestrant in Patients With Previously Treated ER-positive, HER2-negative Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study to Evaluate D-0502 in Subjects With ER+ Her2- Locally Advanced or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0502-303
Record Dates: First submitted 2024-12-20; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- D-0502 (Experimental)
  Interventions: Drug: D-0502
- Fulvestrant (Active Comparator)
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: D-0502 — * Dosage form: Tablet
  * Administration route: Oral, once a day
  Arms: D-0502
Drug: Fulvestrant — * Dosage form: Injection
  * Administration route: Intramuscular injection, once a month, and another dose administered two weeks after the first dose
  Arms: Fulvestrant

SUMMARY:
This is a randomized, parallel-controlled, open-label, multicenter clinical study to assess the efficacy and safety of D-0502 in the treatment of subjects with ER-positive, HER2-negative locally advanced or metastatic breast cancer with fulvestrant injection as a control drug.

ELIGIBILITY:
Inclusion Criteria:

* Subjects pathologically confirmed with ER-positive, HER2-negative breast cancer;
* Subjects with locally advanced (unresectable) or metastatic breast cancer who have disease recurrence during or after adjuvant endocrine therapy, or whose disease has progressed after 1-2 lines of systemic endocrine therapy;
* Presence of at least 1 measurable lesion that can be measured by CT or MRI based on RECIST V1.1 criteria; in the absence of measurable lesions, subjects with evaluable bone lesions [osteolytic or mixed (osteolytic + osteogenic) bone lesions] are also acceptable. Lesions that have been previously treated with radiotherapy or other local therapy can be regarded as measurable lesions only if there is disease progression as confirmed by imaging examination;
* Expected survival time ≥ 12 weeks;

Exclusion Criteria:

* Subjects with unstable or symptomatic or progressive central nervous system (CNS) metastases. Subjects with a history of brain metastases who are clinically stable and have no CNS disease progression confirmed by brain MRI or CT (if MRI is not appropriate) can be enrolled (MRI or CT examination must be conducted at least 4 weeks after the last brain radiotherapy);
* Subjects with locally advanced or metastatic breast cancer who have previously received more than 2 prior systemic chemotherapy;
* Subjects are unsuitable for endocrine therapy judged by the investigator, including uncontrolled pleural effusion, ascites or pericardial effusion;
* Subjects with concomitant medical conditions that the investigator believes may increase the risk of toxicity, such as serious cardiovascular, respiratory or neurological diseases;
* Prior treatment with a selective estrogen receptor degrader (SERD)/selective estrogen receptor covalent antagonist (SERCA), such as fulvestrant, GDC-9545, AZD9833, SAR-439859, Zn -c5, LX-039, HS234, etc.;
* Pregnant or lactating females;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) assessed by Independent Review Committee (IRC) | From enrollment to the end of treatment, up to 2 years

SECONDARY OUTCOMES:
Progression free survival (PFS) -assessed by investigators | From enrollment to the end of treatment, up to 2 years
Objective response rate (ORR) -assessed by IRC and investigators | From enrollment to the end of treatment, up to 2 years
Clinical benefit rate (CBR) -assessed by IRC and investigators | From enrollment to the end of treatment, up to 2 years
Disease control rate (DCR)-assessed by IRC and investigators | From enrollment to the end of treatment, up to 2 years
Clearance (Cl) of D-0502 | on Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1 (each cycle is 28 days)
Overall Survival (OS) | From end of treatment to end of study, about 2 years
Number of participants with adverse events/serious adverse events and abnormal laboratory test results | From enrollment to 30 days after last dose
Volume of distribution (Vd) of D-0502 | on Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, Principal Investigator — Cancer Hospital; Qingyuan Zhang, MD, Principal Investigator — Harbin
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang